CLINICAL TRIAL: NCT06693362
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Safety and Efficacy of Uterine Blood Mesenchymal Stem Cells (SC01009) Injection for the Treatment of Severe Pneumonia Caused by Viruses
Brief Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Safety and Efficacy of Uterine Blood Mesenchymal Stem Cells Injection for the Treatment of Severe Pneumonia Caused by Viruses
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shulan (Hangzhou) Hospital (Other); Shulan(Quzhou) Hospital (Unknown); West China Hospital (Other); Zhejiang University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Shanghai Zhongshan Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZJSCHZ-SC01009-01; CTR20243748 (Other: China drug trials)
Record Dates: First submitted 2024-11-08; First posted 2024-11-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Severe Viral Pneumonia(Not Include COVID-19)
Keywords: severe pneumonia; Safety and Efficacy; Uterine blood mesenchymal stem cells; cell therapy; Phase I clinical trial
MeSH Terms: conditions — Pneumonia | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Control Group (Placebo Comparator): Received SC01009 placebo plus standard treatment
  Interventions: Drug: Placebo; Other: Standard Treatment
- The Treatment Group (Experimental): Received SC01009 in addition to standard treatment.
  Interventions: Drug: Drug therapy; Other: Standard Treatment

INTERVENTIONS:
Drug: Placebo — The Menstrual blood derived mesenchymal stem cells（Men-MSCs）Placebo is administered via intravenous infusion, divided into 3 separate infusions, conducted on alternate days (i.e., Day 1, Day 3, and Day 5).The placebo must be thawed, and 3 vials of placebo must be diluted into 500ml of compound electrolyte injection solution. The medication is administered via intravenous infusion, starting with a slow drip for the first 15 minutes (30-40 drops per minute), and completed within 120 minutes to ensure cell viability. During the infusion process, the infusion bag can be gently shaken appropriately to ensure even suspension of the cells.
  Arms: The Control Group
Drug: Drug therapy — The Menstrual blood derived mesenchymal stem cells（Men-MSCs) injection (SC01009) is administered via intravenous infusion, with a total dose of 9×10^7 cells, divided into 3 separate infusions, conducted on alternate days (i.e., Day 1, Day 3, and Day 5), with each infusion consisting of 3×10^7 cells.Before the infusion, SC01009 injection must be thawed, and 3 vials of SC01009 must be diluted into 500ml of compound electrolyte injection solution. The medication is administered via intravenous infusion, starting with a slow drip for the first 15 minutes (30-40 drops per minute), and completed within 120 minutes to ensure cell viability. During the infusion process, the infusion bag can be gently shaken appropriately to ensure even suspension of the cells.
  Arms: The Treatment Group
Other: Standard Treatment — Anti-infective and anti-inflammatory drugs: For hospitalized patients with CAP, it is recommended to use β-lactams alone or in combination with doxycycline, minocycline, macrolides, or respiratory quinolones alone.
  Corticosteroids: For patients with septic shock, hydrocortisone hemisuccinate 200 mg/day is recommended. The medication should be discontinued promptly after the correction of septic shock, and the duration of use should generally not exceed 7 days.
  Antiviral drugs: Oseltamivir, acyclovir, etc.
  Antipyretic drugs for those with high fever: such as aspirin, acetaminophen, indomethacin, sulindac, naproxen, etc.
  Cough and expectorant drugs for cough and phlegm: ambroxol hydrochloride, acetylcysteine tablets, bromhexine, nacetylethylenediamine, pentedonate, etc.
  Low molecular weight heparin: For elderly hospitalized CAP patients, the risk of deep vein thrombosis should be assessed, and low molecular weight heparin should be applied for prevention when necessary.

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the safety and efficacy of Menstrual blood-derived Mesenchymal Stem Cells (SC01009) injection for the treatment of severe pneumonia caused by viruses. The purpose of the study is to assess the safety and efficacy of SC01009 injection in combination with standard treatment in patients with severe pneumonia caused by viruses. Viral pneumonia refers to acute inflammation of the lung parenchyma and/or interstitium caused by viral infections, which often leads to varying degrees of hypoxia and infection symptoms in the body, typically manifesting as fever, cough, wheezing, shortness of breath, and moist rales in the lungs, along with abnormalities in chest imaging [such as X-rays, computed tomography (CT), etc.]. Viral severe pneumonia is aggressive in onset, initially presenting with fever, cough, and rhinorrhea; it then rapidly progresses to severe toxic symptoms, with respiratory manifestations including cough and dyspnea, producing white mucoid sputum, purulent sputum, or pink frothy sputum. Severely ill patients are often in a critical state of life, endangering the patient's circulatory system and being in a state of respiratory failure requiring ventilator support. Active treatment of viral severe pneumonia, with appropriate measures, can lead to complete recovery of pulmonary function. If respiratory failure or poor circulatory function occurs and ultimately cannot be corrected, the prognosis is poor. Viral severe pneumonia follows clinical pathways (antiviral treatment guidelines and antiviral drug instructions) for antiviral treatment and appropriate adjunctive therapy. Mesenchymal stem cells (MSCs) are a type of multipotent stem cell with the potential for self-renewal and differentiation, characterized by self-renewal, multilineage differentiation, low immunogenicity, and paracrine functions, capable of homing to damaged areas, promoting epithelial tissue repair, suppressing inflammation, and inhibiting abnormal proliferation of fibroblasts.

SC01009 injection is a cellular therapy product developed by Zhejiang Shengchuang Precision Medical Technology Co., Ltd., with its active ingredient being Menstrual blood-derived Mesenchymal Stem Cells (Men-MSCs). Men-MSCs are derived from allogeneic endometrial tissue of women, and preclinical studies have shown that SC01009 is safe and effective in animals, supporting further clinical development.

DETAILED DESCRIPTION:
Severe Pneumonia Caused by Viruses: This includes, but is not limited to, severe pneumonia caused by infections such as respiratory syncytial virus, influenza virus, rhinovirus, human metapneumovirus, adenovirus, etc.; coronavirus is excluded. Diagnostic Criteria: Subjects with pneumonia caused by viral infections. According to the diagnostic criteria for adult community-acquired pneumonia (CAP) in China's 2018 primary care guidelines, a diagnosis of severe pneumonia can be made if one of the following main criteria or at least three secondary criteria are met. Main criteria: ① Need for endotracheal intubation for mechanical ventilation; ② Septic shock requiring vasopressors despite aggressive fluid resuscitation. Secondary criteria: ① Respiratory rate ≥30 breaths/min; ② Oxygenation index ≤250 mmHg (1 mmHg = 0.133 kPa); ③ Multilobar infiltrates; ④ Altered mental status and/or disorientation; ⑤ Blood urea nitrogen ≥7.14 mmol/L; ⑥ Systolic blood pressure <90 mmHg requiring aggressive fluid resuscitation. Viral Detection Methods: The type or subtype of infecting virus is confirmed by nucleic acid testing of patient samples (oropharyngeal swabs, nasopharyngeal swabs, nasopharyngeal aspirates, tracheal aspirates, sputum, and other respiratory specimens, blood samples). Severe pneumonia (SP) is a serious respiratory disease that has emerged globally in recent years, with complex pathogenesis and difficult treatment. Due to different causes, different pathogens, and different situations leading to lung tissue (bronchioles, alveoli, interstitium) inflammation, there are similar or identical pathophysiological processes. When they develop to a certain stage of the disease, they can all worsen and become SP, causing organ dysfunction or even threatening life . SP is associated with high mortality (short-term and long-term) and pulmonary and extrapulmonary complications. Proper diagnosis and early initiation of adequate antimicrobial treatment for patients with severe pneumonia are key to improving the survival rate of critically ill patients. Viral pneumonia is an acute inflammation of the terminal airways, alveolar cavities, and/or interstitium of the lungs caused by viral infections, often resulting from the downward spread of upper respiratory tract infections. It is more common in winter and spring, and can be sporadic, epidemic, or explosive. Viral pneumonia often causes varying degrees of hypoxia and infection symptoms in the body, usually manifesting as fever, cough, wheezing, shortness of breath, and moist rales in the lungs, along with abnormalities in chest imaging [such as X-rays, computed tomography (CT), etc.]. Common pathogens include influenza A virus, parainfluenza virus, adenovirus, coronavirus, coxsackievirus, cytomegalovirus, respiratory syncytial virus, measles virus, varicella virus, etc. The imaging manifestations of viral pneumonia are diverse, but the lesions are often multiple and diffuse, distributed along the periphery and around bronchovascular bundles, with early presentations of multiple small patchy shadows and interstitial changes, thickening of the interlobular and intralobular septa; as the disease worsens, it manifests as multiple ground-glass opacities, which can progress to patchy, nodular, or large confluent consolidations . Typically, viruses from the same virus family have similar pathogenic mechanisms, hence the imaging of viral pneumonia they cause is similar. In terms of pathological characteristics, different severe viral pneumonias also share commonalities . The main manifestations are histological patterns of acute interstitial pneumonia changes, with or without diffuse alveolar damage. Grossly: Lung tissue is enlarged in volume and increased in weight due to congestion and edema (varying with the degree of lesions), with hemorrhagic areas appearing purplish red, and milder lesions may not be apparent. Microscopically: The lesions can be roughly divided into early, middle, late, and terminal stages. Viral severe pneumonia is aggressive in onset, initially presenting with fever, cough, and rhinorrhea; it then rapidly progresses to severe toxic symptoms, with respiratory manifestations including cough and dyspnea, producing white mucoid sputum, purulent sputum, or pink frothy sputum. Wheezing is a significant feature that distinguishes viral pneumonia from bacterial pneumonia, often accompanied by shortness of breath and fever, with severe cases potentially exhibiting lower chest wall inspiratory retractions, perioral cyanosis, and nasal flaring. Physical examination of the lungs often reveals fine to medium moist rales and expiratory wheezing sounds. Chest X-rays may show interstitial infiltrates, patchy shadows, and increased transparency in both lungs, with potential atelectasis. Peripheral blood white blood cell counts are mostly normal, with neutrophil proportions not high, and in cases of bacterial coinfection, white blood cell and neutrophil counts increase. C-reactive protein (CRP) can be normal or slightly elevated. Severely ill patients are often in a critical state of life, endangering the patient's circulatory system, and are in a state of respiratory failure requiring ventilator support. Active treatment of viral severe pneumonia, with appropriate measures, can lead to complete recovery of pulmonary function. If respiratory failure or poor circulatory function occurs and ultimately cannot be corrected, the prognosis is poor. In recent years, new viruses such as the H1N1 influenza virus, H7N9 avian influenza virus, SARS coronavirus (SARS CoV), and Middle East respiratory syndrome coronavirus (MERS-CoV) have emerged as new public health issues, leading to outbreaks or epidemics of viral pneumonia on a global or regional scale.

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following criteria to be eligible for this trial:

1. Aged between 18 and 85 years, regardless of gender;
2. Meet the 2018 primary care diagnostic criteria for severe community-acquired pneumonia (CAP) in adults in China; (Diagnosed according to the diagnostic criteria in the "2018 Guidelines for the Diagnosis and Treatment of Community-Acquired Pneumonia in Adults in Primary Care in China." Severe pneumonia can be diagnosed with one of the following major criteria or ≥3 minor criteria. Major criteria: ① Requires endotracheal intubation for mechanical ventilation; ② Septic shock requiring vasoactive medication after aggressive fluid resuscitation. Minor criteria: ① Respiratory rate ≥30 breaths/min; ② Oxygenation index ≤250 mmHg (1 mmHg=0.133 kPa); ③ Multilobar infiltrates; ④ Altered consciousness and/or disorientation; ⑤ Blood urea nitrogen ≥7.14 mmol/L; ⑥ Systolic blood pressure requiring aggressive fluid resuscitation.)
3. Viral infection confirmed by nucleic acid testing from patient specimens (oropharyngeal swabs, nasopharyngeal swabs, nasopharyngeal aspirates, tracheal aspirates, sputum, and other respiratory specimens, blood specimens), excluding SARS-CoV-2;
4. Compliance with the policies and institutional arrangements for pathogen control by the Health Commission of the region (country) where the experimental center is located;
5. Voluntarily sign and provide written informed consent.

Exclusion Criteria: • Patients who meet any of the following criteria are not eligible for this trial:

1. Clearly diagnosed infections caused by non-viral pathogens, including tuberculosis, bacterial pneumonia, mycoplasma pneumonia, chlamydial pneumonia, or other atypical pathogens causing pneumonia, as defined in the "Clinical Laboratory Manual";
2. Severe pneumonia of unknown viral infection, i.e., the viral pathogen infecting the patient is not well documented and recognized in current literature;
3. History of cancer or clinical examination confirming premalignant lesions at screening;
4. Use of extracorporeal membrane oxygenation (ECMO) at screening;
5. History of acute cerebral infarction within 3 months before screening, or history of deep vein thrombosis or pulmonary embolism at screening;
6. Active immunosuppression including: a) Chemotherapy within the last 4 weeks; B) Continuous use of corticosteroid treatment (equivalent to prednisone ≥1mg/kg·d) for nearly 4 weeks; C) Treatment with immunosuppressants (cyclophosphamide, azathioprine, methotrexate, cyclosporin) within 4 weeks; d) Absolute neutrophil count <0.5×10^9/L;
7. Severe cardiovascular disease within 6 months before screening, including unstable heart disease, myocardial infarction, NYHA Class III or IV heart failure, complete left bundle branch block, or second or third degree atrioventricular block;
8. Abnormal and clinically significant test results for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, and syphilis treponemal (syphilis) antibody;
9. Severe dysfunction of the liver and kidneys;
10. History of poorly controlled mental illness;
11. Known or suspected allergy to the active or inactive ingredients of the study medication;
12. Pregnant or breastfeeding women and women of childbearing age who are not sterilized/refuse to use medically accepted effective contraception during the study period;
13. Men who are not sterilized/refuse to use medically accepted effective contraception during the study period;
14. Those who have participated in other clinical trials (excluding those who have not taken medication) or who have previously received stem cell therapy;
15. Other circumstances deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE/SAE | from the time of medication on day 1 until 24 weeks ± 7 days after discharge, an average of 2 years.
  Incidence of adverse events/serious adverse events
Infusion reactions | On days D1, D3, and D5, during the infusion and within 8 hours after the completion of the infusion, an average of 10 hours
  Infusion reactions (including fever, rigors, itching, hypotension, dyspnea, chest discomfort, rash, urticaria, angioedema, wheezing, tachycardia, and allergic reactions) during the administration period (approximately 2 hours) and within 8 hours after the completion of the infusion, including the time period from the first dose (start of infusion) to 8 hours after the last dose (given on alternate days for a total of 3 times)
Inflammatory markers | from the time of patient infusion to discharge，an average of 3 months
  White Blood Cell count (WBC), Neutrophil percentage (N%), C-reactive protein (CRP), Procalcitonin (PCT), Interleukin-6 (IL-6), IL-8, IL-10, Tumor Necrosis Factor-alpha (TNF-α), Interferon-alpha (IFN-α), Interferon-gamma (IFN-γ) will be combined as the "Inflammatory markers".
Immune markers | from the time of patient infusion to discharge, an average of 3 months
  Immune markers from the time of patient infusion to discharge: Absolute count of CD3, Absolute count of CD4, Absolute count of CD8, CD4+/CD8+ ratio.
Mortality | 28 days
  The all-cause mortality rate within 28 days after enrollment (the ratio of the total number of deaths from all causes to the total number of subjects).
Pneumonia improvement time | 28 days
  The time required for improvement of severe pneumonia after enrollment.
Pneumonia improvement rate | 28 days
  The improvement rate of pneumonia within 28 days after enrollment

SECONDARY OUTCOMES:
Hospital stay | starting from the day a patient is enrolled in a study or treatment protocol and continues until the day of their discharge from the hospital, an average of 3 months.
  The duration of hospital stay after enrollment
ICU stay | the period commencing from the day a patient is enrolled in a clinical study or treatment protocol and ending on the day the patient is discharged from the intensive care unit (ICU), assessed up to 3 months
  The duration of ICU stay after enrollment
All-cause mortality | 8 weeks
  All-cause mortality of subjects 8 weeks after enrollment
viral pneumonia improvement | 28 days
  The time required for viral pneumonia to improve (improvement is defined as reaching clinical stability after treatment).
ARDS incidence rate | From the time the patient enters the study until they discharge due to death or other reasons，an average of 3 months.
  The incidence of viral pneumonia patients progressing to Acute Respiratory Distress Syndrome (ARDS) during the hospital stay
Ventilator free days | 4 weeks
  The time without ventilator use within 4 weeks after hospitalization following enrollment
SOFA score | From the time the patient enters the study until they exit from the ICU due to death or other reasons，assessed up to 3 months.
  The SOFA (Sequential Organ Failure Assessment) score upon admission to and discharge from the ICU
Chest imaging change | From the time of screening through to the 4-week ± 7 days follow-up period post-hospital discharge, which spans an average of 4 months.
  Chest imaging changes at the time of screening, plus or minus 3 days on Day 7 of the trial period, during discharge visit, and at the 4-week ± 7 days follow-up after hospital discharge
laboratory index | From the time the patient enters the study until they discharge due to death or other reasons，an average of 3 months.
  Serum C-reactive protein (CRP), D-dimer, procalcitonin, and cytokine levels in patients from enrollment to discharge during the infusion period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No